CLINICAL TRIAL: NCT00902759
Title: Fatigue, Physical Functioning, and Quality of Life in Patients With Pancreatic and Periampullary Cancers Following Surgery, Chemotherapy, and/or Radiation Therapy
Brief Title: Fatigue and Pancreas and Bile Duct Cancer Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08D.574; 2008-37 (Other: CCRRC); JT 1371 (Other: JeffTrial Number)
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
Keywords: Surgery; Chemotherapy; Radiation Therapy; Pancreatic cancer; Fatigue
MeSH Terms: conditions — Pancreatic Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Group (No Intervention): Participants randomized to the usual care group will be encouraged to return to their "usual" or pre-surgical levels of activity. Usual care of post-surgical PC and peri-ampullary patients typically includes encouragement to walk and be active as they can be by the surgeons, surgical nurses and the nurse practitioners. Participants in the usual care group will not receive an individual "Exercise Prescription" at the time of entry. The usual care group will perform a baseline walk. Participants in the usual care group will not receive an individual "Exercise Prescription" at the time of entry nor will they will a telephone call every month. Repeat questionnaires will be performed at 6 months.
- Walking Program (Experimental): Participants in the intervention arm will participate in a walking program consisting of a 6 week graduated walking program. There are three phases to the walking program, Phase 1 is Warm-up, Phase 2 is Brisk Walking and Phase 3 is Cool Down. Phase 1 is the same for all 6 weeks, and consists of a slow 5 minute walk. In Months 1 and 2, Phase 2 is a 10 minute brisk walk. In Months 3 and 4, Phase 2 is a 20 minute brisk walk. In Months 5 and 6, Phase 2 is a 25 - 30 minute brisk walk. Phase 3 is the same for all 6 weeks and consists of a 5 minute rest/cool down period.
  Interventions: Other: Walking Program

INTERVENTIONS:
Other: Walking Program — "Brisk" walking is defined as faster than the slow walk, but not to exhaustion and not a running pace. Participants will be instructed to walk at home, at a gym or in a shopping mall for as far as possible on a level surface, wearing appropriate footwear as described in the walking booklet. (Patients may continue to walking longer if they desire and are symptom free). Participants should stop or slow down if they experience any discomfort (such as uncomfortable shortness of breath, chest pain, or body pain). The goal is to eventually walk for 90-120 minutes per week in three to four sessions. Participants will not be asked to take their pulse or to record their perceived exertion in order to simplify the program.
  Arms: Walking Program

SUMMARY:
The purpose of this pilot study is to determine the effects of a walking program on fatigue, physical functioning and QOL in patients with pancreatic and periampullary cancers who have had surgery or are undergoing adjuvant therapy with chemotherapy (CT) and/or radiation therapy (RT). This pilot study will utilize the walking program developed by Mock et al. (2001), in their investigation of the improvement of fatigue and QOL in breast care patients following surgery who were receiving CT, RT or biotherapy. No studies published to date have utilized a progressive walking program in post-operative pancreas and ampullary cancers to determine if it reduces adverse effects, such as fatigue or improves functionality and QOL scores.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is the fourth leading cause of cancer death in men and fifth in women in the US (Jemal, Sigel, Ward, Murray, Xu, Thun et al., 2007). According to the American Cancer Society, the reported incidence of PC is roughly 37,000 cases per year, with approximately 33,000 annual deaths (2007). Periampullary cancers are less common; there were 9,250 incident cancers of the biliary tract in 2007, with 3,250 resultant deaths (Jemal et al., 2007).

Five-year survival rates for untreated PC and periampullary cancers are poor, approximately 4%. Surgery offers the only hope of a cure for these patients. Following resection, the reported median survival is 12-18 months, with a five-year survival of 10-40% for patients with PC (Cleary, Gryfe, Guindi, 2004; Ishikawa, Ohihashi, Yamada, Sasaki, Imaoka, Nakaizumi et al., 2002; Sohn, Yeo, Cameron, Koniarais, Kaushal, Abrams, et al., 2000; & Conlon, Klimstra, & Brennan, 1996) and somewhat higher rates for patients with periampullary cancers. Five-year post-resection survival rates may approach 40% when performed at specialized major medical institutions and when favorable pathologic predictors are identified (Sohn et al.). In recent years, improved post-resection survival is due in part to lower perioperative mortality, and partially due to aggressive resection of early, low stage tumors. Long-term survival is considerably lower when resection is performed at low volume pancreatic surgery institutions and postoperative mortality is significantly higher (Birkmeyer, Siewers, Finlayson, Stukel, Lucas, Batista, et al., 2002).

As patients with pancreatic and periampullary cancers experience improved survival rates and live longer, issues regarding adverse symptoms, physical function and quality of life become more important. Fatigue and pain are commonly reported symptoms in patients undergoing CT and RT, with fatigue the most universally reported symptom (Given, Given, McCorkle, Kozachik, Cimprich, Rahbar, Wojcik, 20002). Fatigue can lead to a decrease in activity levels and in one's overall QOL. Exercise has been found to effectively decrease fatigue levels and improve functional capacity in patients with breast and prostate cancer (Mock, Pickett, Ropka, Lin, Rhodes, McDaniel, et al. 2001; Segal, R., Reid, R., Courneya, K, Malone, S., Parliament, M., Scott, C., et al., 2003; MacVicar, Winningham, & Nickel, 1989).

No study to date has reported on the effects of an exercise program on fatigue levels, physical functioning or QOL in post-operative pancreatic and periampullary cancer patients.

This pilot study will employ a quasi-experimental study design that is prospective in nature and randomizes patients to either the intervention group or the usual care group.

Participants will complete the Piper Fatigue Scale (PFS) and the MOS SF-36 QOL questionnaire post-operatively prior to hospital discharge or at the first office visit, and again at the end of six months or at the conclusion of adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic diagnosis of adenocarcinoma of pancreas or periampullary cancers, Stage I, II, or III
* Treatment included surgery alone, or adjuvant treatment with CT and/or RT
* Men and women ≥ 18 years of age
* Residents of the USA
* Surgery performed at TJUH, Philadelphia, PA
* CT or RT performed at TJUH, Jefferson system affiliate hospital, or elsewhere
* Patients receiving neoadjuvant therapy with CT or RT, or both, who subsequently are re-staged and eligible for surgery

Exclusion Criteria:

* The presence of co-morbidities that would preclude involvement in a walking program (wheelchair bound, severe arthritis, dizziness)
* Primary residence outside the USA
* Medical management alone for pancreas or periampullary cancer (i.e. not a surgical candidate)
* Stage IV (metastatic) cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-01-09 (Actual); Primary Completion 2011-01-07 (Actual); Study Completion 2015-04-15 (Actual)

PRIMARY OUTCOMES:
FACIT (Facit Fatigue Scale) and Medical Outcomes Study Short Form-36 (MOS-SF-36) questionnaires | 6 months
  Questionnaires will be completed after surgery but prior to initiation of chemotherapy (CT) or radiation therapy (RT) and again 6 months after hospital discharge or at the completion of adjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Yeo, PhD, MPH, MSN, AOCNP, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Yeo TP, Burrell SA, Sauter PK, Kennedy EP, Lavu H, Leiby BE, Yeo CJ. A progressive postresection walking program significantly improves fatigue and health-related quality of life in pancreas and periampullary cancer patients. J Am Coll Surg. 2012 Apr;214(4):463-75; discussion 475-7. doi: 10.1016/j.jamcollsurg.2011.12.017. Epub 2012 Feb 7. PMID 22321518
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org